CLINICAL TRIAL: NCT00640965
Title: Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Two-Arm, Multi-Center Phase II Trial to Assess the Safety, Tolerability, and Efficacy of DP-VPA (up to 900 mg) Once Daily for 10 Weeks in Adult Subjects With Migraine
Brief Title: DP-VPA for Migraine Prophylaxis, a Pilot Efficacy Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: STUDY WAS NOT STARTED
Sponsor: D-Pharm Ltd. (Industry)
Responsible Party: Dr. Gilad Rosenberg, D-Pharm Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ptcl-01325
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — DP-VPA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): DP-VPA
  Interventions: Drug: DP-VPA
- B (Placebo Comparator)
  Interventions: Drug: DP-VPA Placebo

INTERVENTIONS:
Drug: DP-VPA — DP-VPA dose escalation to 900mg, then continued for 8 weeks
  Arms: A
Drug: DP-VPA Placebo — Matching Placebo to Active, dose escalation, then continued for 8 weeks
  Arms: B

SUMMARY:
The study will evaluate if DP-VPA, a derivative of valproate (a drug that is commonly used for the prevention of migraine attacks), can reduce the rate of migraine attacks.

Migraine patients will take DP-VPA or placebo (an inactive look-alike drug) every morning and will have to report any migraine attacks they have during the study's 18-week follow up.

DETAILED DESCRIPTION:
The multi-center trial has a double-blind, randomized, placebo-controlled, parallel-group design and will be carried out in Israel. Approximately 40 adult subjects with migraine will be randomly assigned (1:1) to either DP-VPA (maximum of 900mg/day) or placebo. Active and placebo will be administered orally and once-daily on an add-on basis, i.e. other permissible ongoing medications will be continued. Total study duration per subject will be 18 weeks. Subjects will report on their migraine attacks frequency and other attack characteristics using weekly diaries.

ELIGIBILITY:
Inclusion criteria (abridged)

* Male and female subjects with migraine with or without aura fulfilling the diagnostic criteria of the International Classification of Headache Disorders
* 3 to 6 migraine attacks per month
* Concomitant prophylactic migraine treatment with a beta-blocker or amitriptyline that has been stable in the proceeding 3 months. No changes in this concomitant treatment will be allowed until the end of study follow-up.

Exclusion criteria (abridged)Chronic migraine (>15 days of migraine/ month).

* Migraine complicated by medication-overuse headache.
* Allergy or hypersensitivity to valproic acid, valproate sodium, or soy.
* Known contraindications to valproic acid.
* Pregnancy.
* Breastfeeding female subjects.
* Subjects with significant hepatic dysfunction indicated by SGOT or SGPT >3 times the upper limit of normal at screening.
* Renal impairment indicated by serum creatinine >1.5mg/dL at screening.
* Potentially fertile and sexually active women who do not practice reliable contraception.
* Men who do not practice reliable barrier contraception.
* Concomitant use of antipsychotic, antidepressant or antiepileptic therapy - with the exception of amitriptyline - within 1 month of screening, or a medical condition that is likely to require such treatment during the trial participation.
* An active central nervous system disease deemed to be unstable or progressive during the course of the study that may confound the interpretation of the study results.
* Any medical disorder that may makes the subject unlikely to fully complete the study- Blood coagulation disorder.
* Concomitant drugs known to interact with VPA.- Alcohol or other drugs abuse.
* Therapy with another investigational product within 30 days prior start of study.
* Concomitant participation in another trial or study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Migraine attacks frequency | 6 months

SECONDARY OUTCOMES:
Migraine days | 6 months
Responders (subjects with >50% decrease in migraine frequency) | 6 months
Triptan consumption | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Rosenberg, M.D., Study Director — D-Pharm Ltd.
Locations (6):
- Israel (6):
  - Rambam Medical Center, Haifa
  - Bnei Zion Medical Centre, Haifa
  - Wolfson Medical Center, Holon
  - Beilinson Medical Centre, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky